CLINICAL TRIAL: NCT06167421
Title: Comparison of Kimura Versus Warshaw Technique for Laparoscopic Spleen-Preserving Distal Pancreatectomy: A Multicenter Randomized Controlled Clinical Trial
Brief Title: Comparison of Kimura Versus Warshaw Technique for Laparoscopic Spleen-Preserving Distal Pancreatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Qilu Hospital of Shandong University (Other); The Third Affiliated Hospital of Soochow University (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, President of Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPAC-7
Record Dates: First submitted 2023-11-20; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Tumor, Benign; Pancreatic Neuroendocrine Tumor; Solid Pseudopapillary Tumor of the Pancreas
Keywords: Pancreatic benign or low-grade malignant tumors; Minimally invasive spleen-preserving distal pancreatectomy; Kimura technique; Warshaw technique; Prognosis
MeSH Terms: conditions — Pancreatic Neoplasms; Adenoma, Islet Cell

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kimura group (Experimental): Laparoscopic spleen-preserving distal pancreatectomy using the Kimura technique.
  Interventions: Procedure: Laparoscopic spleen-preserving distal pancreatectomy using the Kimura technique
- Warshaw group (Active Comparator): Laparoscopic spleen-preserving distal pancreatectomy using the Warshaw technique.
  Interventions: Procedure: Laparoscopic spleen-preserving distal pancreatectomy using the Warshaw technique

INTERVENTIONS:
Procedure: Laparoscopic spleen-preserving distal pancreatectomy using the Kimura technique — The laparoscopic spleen-preserving distal pancreatectomy using the Kimura technique is defined as a surgical procedure that aims to remove the distal part of the pancreas while preserving the spleen by maintaining the splenic artery and vein (Hepatogastroenterology. 2003;50:2242).
  Arms: Kimura group
Procedure: Laparoscopic spleen-preserving distal pancreatectomy using the Warshaw technique — Warshaw technique laparoscopic spleen-preserving distal pancreatectomy is defined as a surgical procedure that aims to preserve the spleen while removing the distal part of the pancreas. It involves ligating the splenic artery and vein, while preserving the left gastroepiploic artery and short gastric vessels (Arch Surg. 1988;123:550).
  Arms: Warshaw group

SUMMARY:
This study aims to compare the surgical outcomes of laparoscopic spleen-preserving distal pancreatectomy using the Kimura technique versus the Warshaw technique. The primary focus is on the rates of unplanned splenectomy, occurrence of severe complications, as well as intraoperative and perioperative outcomes of both techniques.

DETAILED DESCRIPTION:
For benign and low-grade malignant tumors of the pancreatic body and tail, laparoscopic distal pancreatosplenectomy (LDP) is commonly recommended due to its shorter hospital stay, lower intraoperative blood loss, and comparable complication rates. The DIPLOMA international multicenter clinical trial further established the non-inferiority of minimally invasive techniques in terms of curative resection for resectable pancreatic body and tail cancers.

As the spleen plays a crucial role in immune defense, splenectomy is associated with increased postoperative infection risk, significant increase in platelet count, and thrombosis. Therefore, for benign and low-grade malignant tumors of the pancreatic body and tail, minimally invasive spleen-preserving distal pancreatectomy should be the preferred approach.

The Kimura technique is the most commonly used and favored spleen-preserving distal pancreatectomy technique. It involves the complete preservation of splenic vessels, resulting in fewer postoperative complications. However, it is time-consuming and challenging due to the identification and ligation of numerous small and short vessels entering the pancreatic body and tail to preserve the fragile splenic artery and vein. On the other hand, the Warshaw technique involves segmental resection of splenic vessels and relies on the left gastroepiploic artery and short gastric vessels for splenic perfusion. It is a simpler procedure with less intraoperative blood loss and shorter operative time. However, it carries an increased risk of postoperative splenic infarction, gastric varices, and secondary bleeding.

Although a higher incidence of splenic infarction has been observed with the Warshaw technique, its clinical relevance remains controversial. Reports indicate that approximately 25% of patients undergoing Warshaw procedure show radiological evidence of asymptomatic gastric varices, but during a follow-up period of up to 21 years, no clinically relevant consequences of gastric varices were observed. Most cases of postoperative splenic infarction are transient and do not require specific treatment. Data from a large pan-European retrospective study showed no significant differences in the clinical incidence of splenic infarction (0.6% vs. 1.6%, P = 0.127) and major complication rates (11.5% vs. 14.4%, P = 0.308) between minimally invasive Kimura and Warshaw techniques.

While Kimura and Warshaw techniques demonstrate comparability in most postoperative outcomes, the former appears to have an advantage in reducing the risk of splenic infarction and gastric varices. Some experts propose a "Kimura-first" strategy. However, there is currently no prospective study comparing these two techniques. Therefore, this study has designed a multicenter randomized controlled clinical trial, focusing on the rates of unplanned splenectomy, severe complication occurrence, and intraoperative and perioperative outcomes of laparoscopic spleen-preserving distal pancreatectomy using the Kimura versus the Warshaw technique. Long-term follow-up will assess clinically relevant outcomes such as splenic ischemia, splenic hyperfunction, gastric varices, and postoperative quality of life. This study aims to provide higher-level evidence in the selection of laparoscopic spleen-preserving distal pancreatectomy techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years, regardless of gender.
* Preoperative clinical diagnosis of benign or low-grade malignant pancreatic tumors.
* Meeting the recommended surgical indications as per guidelines.
* Feasibility of imaging assessment for either Kimura or Warshaw technique laparoscopic spleen-preserving distal pancreatectomy.
* Performance status of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) score.
* Willingness to comply with the study treatment plan, follow-up schedule, and other protocol requirements.
* Voluntarily participating in the study and signing an informed consent form.

Exclusion Criteria:

* Body Mass Index (BMI) > 28 kg/m2 (Chinese obesity standard).
* History of blood disorders, acute or chronic pancreatitis, gastrointestinal bleeding, splenic rupture, or gastric varices (preoperative CT indicating curved vessel structures along the gastric wall with a diameter > 5mm).
* History of abdominal surgery.
* Concomitant primary malignant tumors.
* Suspicion of malignancy based on PET-CT or other imaging examinations.
* Severe impairment of cardiac, liver, or kidney function (NYHA class 3-4, ALT and/or AST exceeding three times the upper limit of normal, Creatinine exceeding the upper limit of normal).
* Planned pregnancy or pregnancy and lactating women.
* Participants currently involved in other clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Unplanned splenectomy rate | Immediately after the surgery.
  The unplanned splenectomy rate in both groups will be calculated, and detailed records of the specific reasons will be documented, such as adhesions, bleeding, intraoperative splenic infarction.
Severe complication rate | Within 90 days after surgery.
  The rate of severe complications will be assessed by evaluating the severity of postoperative complications using the Clavien-Dindo classification system. In this classification system, complications graded as III and above are considered severe complications.

SECONDARY OUTCOMES:
Spleen vessel preservation rate | Immediately after the surgery.
  The spleen vessel preservation rate refers to the rate at which the spleen vessels are successfully preserved during surgery. In cases where the Kimura technique is unable to preserve the spleen vessels, salvage Warshaw procedure or splenectomy may be performed. This can include modified Warshaw procedures that involve the simple removal of the splenic artery or splenic vein.
Postoperative Clinically Relevant Spleen Ischemia (CRSI) rate | Through study completion, an average of 3 year.
  CRSI is defined as the occurrence of spleen ischemia requiring splenectomy during either the initial hospitalization or subsequent readmissions. The reasons for the second splenectomy will be recorded.
Postoperative quality of life assessment | Through study completion, an average of 3 year.
  The evaluation will be conducted using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30).
  The EORTC QLQ-C30 is a widely used questionnaire to assess the quality of life. It consists of multiple scales and items that cover various aspects of physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, global health status, and symptom scales.
  Each item in the questionnaire is rated on a four-point Likert scale, ranging from 1 (not at all) to 4 (very much). Some items are reverse-scored, meaning that a higher score indicates a worse outcome. The scores for each scale are then transformed to a 0-100 scale, where a higher score represents a better outcome for functioning scales and a worse outcome for symptom scales.

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, MD, PhD, Principal Investigator — Fudan University

REFERENCES:
- [Background] de Rooij T, van Hilst J, van Santvoort H, Boerma D, van den Boezem P, Daams F, van Dam R, Dejong C, van Duyn E, Dijkgraaf M, van Eijck C, Festen S, Gerhards M, Groot Koerkamp B, de Hingh I, Kazemier G, Klaase J, de Kleine R, van Laarhoven C, Luyer M, Patijn G, Steenvoorde P, Suker M, Abu Hilal M, Busch O, Besselink M; Dutch Pancreatic Cancer Group. Minimally Invasive Versus Open Distal Pancreatectomy (LEOPARD): A Multicenter Patient-blinded Randomized Controlled Trial. Ann Surg. 2019 Jan;269(1):2-9. doi: 10.1097/SLA.0000000000002979. PMID 30080726
- [Background] Asbun HJ, Moekotte AL, Vissers FL, Kunzler F, Cipriani F, Alseidi A, D'Angelica MI, Balduzzi A, Bassi C, Bjornsson B, Boggi U, Callery MP, Del Chiaro M, Coimbra FJ, Conrad C, Cook A, Coppola A, Dervenis C, Dokmak S, Edil BH, Edwin B, Giulianotti PC, Han HS, Hansen PD, van der Heijde N, van Hilst J, Hester CA, Hogg ME, Jarufe N, Jeyarajah DR, Keck T, Kim SC, Khatkov IE, Kokudo N, Kooby DA, Korrel M, de Leon FJ, Lluis N, Lof S, Machado MA, Demartines N, Martinie JB, Merchant NB, Molenaar IQ, Moravek C, Mou YP, Nakamura M, Nealon WH, Palanivelu C, Pessaux P, Pitt HA, Polanco PM, Primrose JN, Rawashdeh A, Sanford DE, Senthilnathan P, Shrikhande SV, Stauffer JA, Takaori K, Talamonti MS, Tang CN, Vollmer CM, Wakabayashi G, Walsh RM, Wang SE, Zinner MJ, Wolfgang CL, Zureikat AH, Zwart MJ, Conlon KC, Kendrick ML, Zeh HJ, Hilal MA, Besselink MG; International Study Group on Minimally Invasive Pancreas Surgery (I-MIPS). The Miami International Evidence-based Guidelines on Minimally Invasive Pancreas Resection. Ann Surg. 2020 Jan;271(1):1-14. doi: 10.1097/SLA.0000000000003590. PMID 31567509
- [Background] Korrel M, Jones LR, van Hilst J, Balzano G, Bjornsson B, Boggi U, Bratlie SO, Busch OR, Butturini G, Capretti G, Casadei R, Edwin B, Emmen AMLH, Esposito A, Falconi M, Groot Koerkamp B, Keck T, de Kleine RHJ, Kleive DB, Kokkola A, Lips DJ, Lof S, Luyer MDP, Manzoni A, Marudanayagam R, de Pastena M, Pecorelli N, Primrose JN, Ricci C, Salvia R, Sandstrom P, Vissers FLIM, Wellner UF, Zerbi A, Dijkgraaf MGW, Besselink MG, Abu Hilal M; European Consortium on Minimally Invasive Pancreatic Surgery (E-MIPS). Minimally invasive versus open distal pancreatectomy for resectable pancreatic cancer (DIPLOMA): an international randomised non-inferiority trial. Lancet Reg Health Eur. 2023 Jul 6;31:100673. doi: 10.1016/j.lanepe.2023.100673. eCollection 2023 Aug. PMID 37457332
- [Background] Casciani F, Trudeau MT, Vollmer CM Jr. Perioperative Immunization for Splenectomy and the Surgeon's Responsibility: A Review. JAMA Surg. 2020 Nov 1;155(11):1068-1077. doi: 10.1001/jamasurg.2020.1463. PMID 32936229
- [Background] Korrel M, Lof S, Al Sarireh B, Bjornsson B, Boggi U, Butturini G, Casadei R, De Pastena M, Esposito A, Fabre JM, Ferrari G, Fteriche FS, Fusai G, Koerkamp BG, Hackert T, D'Hondt M, Jah A, Keck T, Marino MV, Molenaar IQ, Pessaux P, Pietrabissa A, Rosso E, Sahakyan M, Soonawalla Z, Souche FR, White S, Zerbi A, Dokmak S, Edwin B, Hilal MA, Besselink M; European consortium on Minimally Invasive Pancreatic Surgery (E-MIPS). Short-term Outcomes After Spleen-preserving Minimally Invasive Distal Pancreatectomy With or Without Preservation of Splenic Vessels: A Pan-European Retrospective Study in High-volume Centers. Ann Surg. 2023 Jan 1;277(1):e119-e125. doi: 10.1097/SLA.0000000000004963. Epub 2021 Jun 2. PMID 34091515
- [Background] Yongfei H, Javed AA, Burkhart R, Peters NA, Hasanain A, Weiss MJ, Wolfgang CL, He J. Geographical variation and trends in outcomes of laparoscopic spleen-preserving distal pancreatectomy with or without splenic vessel preservation: A meta-analysis. Int J Surg. 2017 Sep;45:47-55. doi: 10.1016/j.ijsu.2017.07.078. Epub 2017 Jul 21. PMID 28735894
- [Background] Warshaw AL. Conservation of the spleen with distal pancreatectomy. Arch Surg. 1988 May;123(5):550-3. doi: 10.1001/archsurg.1988.01400290032004. PMID 3358679
- [Background] Ferrone CR, Konstantinidis IT, Sahani DV, Wargo JA, Fernandez-del Castillo C, Warshaw AL. Twenty-three years of the Warshaw operation for distal pancreatectomy with preservation of the spleen. Ann Surg. 2011 Jun;253(6):1136-9. doi: 10.1097/SLA.0b013e318212c1e2. PMID 21394008
- [Background] Granieri S, Bonomi A, Frassini S, Gjoni E, Germini A, Kersik A, Bracchetti G, Bruno F, Paleino S, Lomaglio L, Frontali A, Cotsoglou C. Kimura's vs Warshaw's technique for spleen preserving distal pancreatectomy: a systematic review and meta-analysis of high-quality studies. HPB (Oxford). 2023 Jun;25(6):614-624. doi: 10.1016/j.hpb.2023.02.009. Epub 2023 Mar 1. PMID 36941150